CLINICAL TRIAL: NCT06232759
Title: Transarterial Chemoembolization Combined With Tyrosine Kinase Inhibitors and Tislelizumab in Unresectable Hepatocellular Carcinoma
Brief Title: TACE Combined With Tyrosine Kinase Inhibitors and Tislelizumab in Unresectable Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Principal Investigator, Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRONT-2
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Tyrosine Kinase Inhibitors; tislelizumab

STUDY DESIGN:
Intervention Model Description: Patients with unresectable hepatocellular carcinoma were received transarterial chemoembolization combined with Tyrosine Kinase Inhibitors and Tislelizumab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transarterial chemoembolization combined with Tyrosine Kinase Inhibitors and Tislelizumab (Experimental): Patients with unresectable hepatocellular carcinoma were received transarterial chemoembolization combined with Tyrosine Kinase Inhibitors and Tislelizumab
  Interventions: Drug: Transarterial chemoembolization combined with Tyrosine Kinase Inhibitors and Tislelizumab

INTERVENTIONS:
Drug: Transarterial chemoembolization combined with Tyrosine Kinase Inhibitors and Tislelizumab — Patients with unresectable hepatocellular carcinoma were received transarterial chemoembolization combined with Tyrosine Kinase Inhibitors and Tislelizumab

SUMMARY:
Most hepatocellular carcinoma (HCC) are found in the intermediate or advanced stage. The patients lose the opportunity of curative surgical resection. In clinical practice, unresectable HCC is often encountered with large tumor lesions and insufficient remaining liver volume. It is expected that the benefit of direct surgical resection will not exceed that of non-surgical treatment if the tumor is limited in scope but with unclear boundaries, surrounding small foci, or adjacent to important vascular structures, or combined with secondary or higher portal vein tumor thrombus. These patients account for a significant proportion of unresectable HCC, but have the potential for surgical resection. If the investigators can make full use of the existing HCC treatment, the patients hope to obtain radical surgical resection opportunities and better long-term survival after tumor shrinkage and tumor necrosis boundary becomes clear.

Transcatheter arterial chemoembolization (TACE) has been the standard arterial treatment for advanced HCC. Tyrosine kinase Inhibitor is the first-line treatment for hepatocellular carcinoma. Tislelizumab is an immune checkpoint inhibitor and a first-line treatment for HCC. This study investigated the efficacy and safety of TACE combined with Tyrosine Kinase Inhibitors and tislelizumab in the treatment of unresectable HCC.

ELIGIBILITY:
Inclusion Criteria:

* Had Child-Pugh score 5-7 liver function, an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, and adequate organ function at the time of treatment initiation;
* With stage Ⅰb, Ⅱa, Ⅱb or Ⅲa hepatocellular carcinoma (HCC) based on the Chinese liver Cancer Staging System (CNLC);
* With unresectable HCC because of insufficient residual liver volume;
* Expected survival time ≥6 months;
* Hematology indexes should meet the following conditions: hemoglobin ≥90 g/L; platelet ≥80; total bilirubin ≤1.5×ULN; alanine transaminase ≤3×ULN; aspertate aminotransferase ≤ 3 x ULN; alkaline phosphatase ≤2.5×ULN; serum albumin ≥28 g/L; serum creatinine ≤1.5×ULN;
* Urinary protein <2+ or 24 h urinary protein quantity < 1.0g;
* For women of reproductive age, contraceptive measures (such as intrauterine devices, contraceptive tablets or condoms) are required during the clinical trial until 120 days after the end of the clinical trial; Women of childbearing age had negative serum or urine HCG test results within 7 days prior to inclusion in the study; For male patients whose partners have reproductive potential, effective contraception should be used during the study period and for 120 days after the end of the study.

Exclusion Criteria:

* Combined with other malignant tumors;
* Previously received local treatment of HCC such as Hepatic Artery Infusion Chemotherapy, transarterial (chemo)embolization, or local ablation;
* Those who have received or are using one of the following three types of drugs in the past 6 months: Immune checkpoint inhibitors, including but not limited to Atezolizumab, Nivolumab, pembrolizumab, Camrelizumab, Tislelizumab, triplizumab, sintilimab, etc.; Molecular targeted therapy, including but not limited to sorafenib, lenvatinib, donafenib, apatinib, regorafenib, anrotinib, bevacizumab, etc.; systemic chemotherapy drugs (such as doxorubicin, oxaliplatin, 5-FU, S-1, etc.);
* The presence of congenital or acquired immunodeficiency diseases (such as HIV positive);
* Active infection, or body temperature ≥ 38.5℃ 7 days before enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | One year
  The proportion of progression-free survival in one year

SECONDARY OUTCOMES:
Overall survival | One year
  The proportion of overall survival in one year

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Ping Liu, M.D, Principal Investigator — The Eighth Affiliated hospital of the Guangxi Medical University
Locations (1):
- Jian-Hong Zhong, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: Yes
Original data can be obtained from the corresponding authors in accordance with privacy/ethical restrictions.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the full paper was published.
Access Criteria: use the data for further analysis, for example, meta-analysis.

REFERENCES:
- [Background] Chen K, Wei W, Liu L, Deng ZJ, Li L, Liang XM, Guo PP, Qi LN, Zhang ZM, Gong WF, Huang S, Yuan WP, Ma L, Xiang BD, Li LQ, Zhong JH. Lenvatinib with or without immune checkpoint inhibitors for patients with unresectable hepatocellular carcinoma in real-world clinical practice. Cancer Immunol Immunother. 2022 May;71(5):1063-1074. doi: 10.1007/s00262-021-03060-w. Epub 2021 Sep 24. PMID 34559308
- [Background] Cheng AL, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Lim HY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Ma N, Nicholas A, Wang Y, Li L, Zhu AX, Finn RS. Updated efficacy and safety data from IMbrave150: Atezolizumab plus bevacizumab vs. sorafenib for unresectable hepatocellular carcinoma. J Hepatol. 2022 Apr;76(4):862-873. doi: 10.1016/j.jhep.2021.11.030. Epub 2021 Dec 11. PMID 34902530
- [Background] Qin S, Kudo M, Meyer T, Bai Y, Guo Y, Meng Z, Satoh T, Marino D, Assenat E, Li S, Chen Y, Boisserie F, Abdrashitov R, Finn RS, Vogel A, Zhu AX. Tislelizumab vs Sorafenib as First-Line Treatment for Unresectable Hepatocellular Carcinoma: A Phase 3 Randomized Clinical Trial. JAMA Oncol. 2023 Dec 1;9(12):1651-1659. doi: 10.1001/jamaoncol.2023.4003. PMID 37796513
- [Background] Qin S, Bi F, Gu S, Bai Y, Chen Z, Wang Z, Ying J, Lu Y, Meng Z, Pan H, Yang P, Zhang H, Chen X, Xu A, Cui C, Zhu B, Wu J, Xin X, Wang J, Shan J, Chen J, Zheng Z, Xu L, Wen X, You Z, Ren Z, Liu X, Qiu M, Wu L, Chen F. Donafenib Versus Sorafenib in First-Line Treatment of Unresectable or Metastatic Hepatocellular Carcinoma: A Randomized, Open-Label, Parallel-Controlled Phase II-III Trial. J Clin Oncol. 2021 Sep 20;39(27):3002-3011. doi: 10.1200/JCO.21.00163. Epub 2021 Jun 29. PMID 34185551